CLINICAL TRIAL: NCT03011450
Title: A Phase 3, Multi-Center, Placebo-Controlled, Randomized, Double--Blind, 12-Week Study With a 40-Week, Active-Controlled, Open-Label Extension to Evaluate the Efficacy and Safety of K-877 in Adult Patients With Fasting Triglyceride Levels ≥500 mg/dL and <2000 mg/dL and Mild or Moderate Renal Impairment
Brief Title: Study to Evaluate the Efficacy and Safety of K-877 in Adult Patients With Fasting High Triglyceride Levels and Mild or Moderate Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K-877-303
Record Dates: First submitted 2016-12-20; First posted 2017-01-05 (Estimated); Results first posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-09

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — K-877 compound; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 12 Week Efficacy (Placebo Comparator): K-877 or placebo comparator for 12 weeks
  Interventions: Drug: K-877; Drug: Placebo (for K-877)
- 40 week extension (Active Comparator): K-877 or fenofibrate comparator for 40 weeks
  Interventions: Drug: K-877; Drug: Fenofibrate

INTERVENTIONS:
Drug: K-877
Drug: Fenofibrate
  Arms: 40 week extension
Drug: Placebo (for K-877)
  Arms: 12 Week Efficacy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of K-877 in adult patients With Fasting High Triglyceride Levels ≥500 mg/dL and <2000 mg/dL and Mild or Moderate Renal Impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to comply with all study requirements and procedures throughout the duration of the study and give written informed consent;
2. Aged ≥18 years;
3. Patients receiving moderate- or high-intensity statin therapy must meet one of the following criteria¹ unless they have any exceptional conditions (see inclusion criterion 4):

   1. Aged ≥21 years with clinical atherosclerotic cardiovascular disease (ASCVD) (history of acute coronary syndrome or myocardial infarction, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack [TIA] presumed to be of atherosclerotic origin, or peripheral arterial disease or revascularization), on a high-intensity statin (or moderate-intensity statin if not a candidate for high-intensity statin due to safety concerns);
   2. Aged ≥21 years with a history of LDL-C ≥190 mg/dL, which is not due to secondary modifiable causes, on a high-intensity statin (or moderate-intensity statin if not a candidate for high-intensity statin due to safety concerns);
   3. Aged 40 to 75 years, inclusive, without clinical ASCVD but with diabetes and a history of LDL-C of 70 to 189 mg/dL, inclusive, on a moderate- or high-intensity statin; or
   4. Aged 40 to 75 years, inclusive, without clinical ASCVD or diabetes, with a history of LDL-C of 70 to 189 mg/dL, inclusive, with estimated 10-year risk for ASCVD of ≥7.5% by the Pooled Cohort Equation on a moderate- or high-intensity statin;
4. Patients currently on a low-intensity statin or not on a statin, must meet one of the following criteria;

   1. Patient does not meet any criteria for moderate- or high-intensity statin therapy listed above (see inclusion criteria, 3.a. through 3.d.);
   2. Patient does meet one or more criteria for moderate- or high-intensity statin therapy listed above (see inclusion criteria 3.a. through 3.d.); but the patient is not a candidate for moderate or high-intensity statin due to safety concerns, or due to partial or complete statin intolerance; or
   3. Patient does meet one or more criteria for moderate- or high intensity statin therapy listed above (see inclusion criteria 3.b. through 3.d., except for 3.a.); but the patient is not a candidate for moderate or high intensity statin for primary prevention after considering individual risk evaluation (e.g. current LDL C ≤70mg/dL) and patient preference;
5. Fasting TG levels ≥500 mg/dL (5.65 mmol/L) and <2000 mg/dL (22.60 mmol/L) based on the mean of Visit 2 (Week -2) and Visit 3 (Week -1).

   * Mild to moderate renal impairment eGFR >= 30mL/min/1.73 and < 90 mL/min/1.73 at Visit 1

Exclusion Criteria:

1. Patients who will require lipid-altering treatments other than study drugs (K-877 or fenofibrate), statins, ezetimibe, or PCSK9 inhibitors during the course of the study. These include bile acid sequestrants, non-study fibrates, niacin (>100 mg/day), omega-3 fatty acids (>1000 mg/day), or any supplements used to alter lipid metabolism including, but not limited to, red rice yeast supplements, garlic supplements, soy isoflavone supplements, sterol/stanol products, or policosanols;
2. Body mass index (BMI) >45 kg/m2 at Visit 1 (Week -8 or Week -6);
3. Patients with type 1 diabetes mellitus;
4. Patients with newly diagnosed (within 3 months prior to Visit 2 [Week -2]) or poorly controlled type 2 diabetes mellitus (T2DM), defined as hemoglobin A1c >9.5% at Visit 1 (Week -8 or Week -6);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2016-11-26 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (240):
- United States (128):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Central Alabama Research, Birmingham, Alabama
  - Cahaba Research, Inc., Birmingham, Alabama
  - Boyett Health Services Inc, Hamilton, Alabama
  - Longwood Research - Saadat Ansari, MD, LLC, Huntsville, Alabama
  - Terence T. Hart, MD, Tuscumbia, Alabama
  - Arrowhead Health Centers, Glendale, Arizona
  - Phoenix Medical Research Institute, LLC, Peoria, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - Clinical Research Institute of Arizona, LLC, Surprise, Arizona
  - iResearch, Little Rock, Arkansas
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Downtown L.A. Research Center, Inc., Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Pacific Coast Cardiology and Research, Newport Beach, California
  - Lucita M. Cruz, MD., Inc., Norwalk, California
  - Integrated Research Center, San Diego, California
  - Optimus Medical Group, San Francisco, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Atlantic Clinical Research Collaborative, Boynton Beach, Florida
  - ALL Medical Research, LLC, Cooper City, Florida
  - S & W Clinical Research, Fort Lauderdale, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - AMPM Research Clinic, Miami Gardens, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - South Florida Research Solutions LLC., Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Meridien Research - Tampa, Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Columbus Regional Health, Columbus, Georgia
  - iResearch, Decatur, Georgia
  - Physicians Research Associates, Inc, Lawrenceville, Georgia
  - Georgia Institute for Clinical Research, Marietta, Georgia
  - Endocrine Research Solutions, Inc, Roswell, Georgia
  - Meridian Clinical Research - Savannah, GA, Savannah, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Lemah Creek Clinical Research, Burr Ridge, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Apex Medical Research, Chicago, Illinois
  - Koch Family Medicine, Morton, Illinois
  - Community Hospital of Anderson and Madison County, Inc, Anderson, Indiana
  - American Health Network - Avon Clinical Research Department, Avon, Indiana
  - Medisphere Medical Research Center, Evansville, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - The Iowa Clinic - Cardiovascular Services, West Des Moines, Iowa
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Research Integrity LLC, Owensboro, Kentucky
  - Clinical Trials Management, LLC - Northshore, Covington, Louisiana
  - Clinical Trials Management LLC - Southshore, Metairie, Louisiana
  - Grace Research, LLC, Shreveport, Louisiana
  - Clinical Trials of America, LLC, West Monroe, Louisiana
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Regeneris Medical, North Attleboro, Massachusetts
  - Aa Mrc, Llc, Flint, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - David M. Headley, MD P.A., Port Gibson, Mississippi
  - Consult and Research Associates, St Louis, Missouri
  - Advance Clinical Research, Inc, St Louis, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Desert Endocrinology Clinical Research Center, Henderson, Nevada
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Lakeshore Primary Care Associate, Hamburg, New York
  - Mid-Hudson Medical Research, PLLC - Hopewell Junction, New Windsor, New York
  - Mid-Hudson Medical Research, PLLC - New Windsor, New Windsor, New York
  - Orchard Park Family Practice, Orchard Park, New York
  - Diabetes and Endocrinology Consultants, P.C., Morehead City, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Sterling Research Group, Ltd. - Auburn, Cincinnati, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Alpha Research Associates, LLC, Dayton, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Ohio Clinical Research - Lyndhurst, Lyndhurst, Ohio
  - Rama Research LLC, Marion, Ohio
  - RAS Health Ltd, Marion, Ohio
  - Summit Research Group, LLC, Munroe Falls, Ohio
  - Ohio Clinical Research, LLC - Willoughby Hills, Willoughby Hills, Ohio
  - COR Clinical Research, LLC., Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Clinical Research Associates of Central PA, LLC, Altoona, Pennsylvania
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Richard M.Kastelic MD and Associates, Johnstown, Pennsylvania
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Center for Medical Research, LLC, Providence, Rhode Island
  - MD First Research, Anderson, South Carolina
  - MDFirst Research - Anderson, Anderson, South Carolina
  - DeGarmo Institute Of Medical Research, Greer, South Carolina
  - MD First Research, Lancaster, South Carolina
  - Family Medicine of SayeBrook, Myrtle Beach, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - PMG Research of Bristol, LLC - State, Bristol, Tennessee
  - Chattanooga Research & Medicine, PLLC, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - Clinical Research Solutions - Smyrna, TN, Smyrna, Tennessee
  - Health Innovation Research Group, Arlington, Texas
  - DCT-AACT, LLC, dba Discovery Clinical Trials, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - Padre Coast Clinical Research, Corpus Christi, Texas
  - Protenium Clinical Research, LLC - Dallas, Dallas, Texas
  - VA North Texas Health Care System - Dallas VA Medical Center (DVAMC), Dallas, Texas
  - Academy of Diabetes, Thyroid and Endocrine, P.A., El Paso, Texas
  - Juno Research, LLC, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Pioneer Research Solutions Inc., Houston, Texas
  - Grace Research, LLC, Huntsville, Texas
  - Protenium Clinical Research, LLC, Hurst, Texas
  - Juno Research, LLC, Katy, Texas
  - FMC Science, Lampasas, Texas
  - Pinnacle Clinical Research, Live Oak, Texas
  - DCT - McAllen Primary Care, LLC, McAllen, Texas
  - San Antonio Premier Internal Medicine, San Antonio, Texas
  - Physician PrimeCare Research Institute, PLLC dba Health Texas Research Institute, San Antonio, Texas
  - Bandera Family HealthCare Research, LLC (BFHC), San Antonio, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - Cardiovascular Associates, Ltd, Virginia Beach, Virginia
  - Exemplar Research Inc. - Fairmont, WV, Morgantown, West Virginia
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin
- Belarus (11):
  - Brest Regional Hospital, Brest
  - Grodno University Hospital, Grodno
  - Gomel Regional Clinical Hospital, Homyel
  - Gomel Regional Clinical Center of Cardiology, Homyel
  - City Clinical Hospital #1, Minsk
  - City Clinical Hospital #9, Minsk
  - Minsk Scientific and Practice Center of Surgery, Transplantology and Hematology, Minsk
  - City Clinical Hospital #10, Minsk
  - Minsk Regional Clinical Hospital, Minsk
  - Mogilev Regional Medical and Diagnostic Center, Mogilev
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Bulgaria (9):
  - Medical Center Diamedical 2013 OOD, Dimitrovgrad
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski EAD- First Cardiology Clinic, Pleven
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski EAD- Second Cardiology Clinic, Pleven
  - University Multiprofile Hospital for Active Treatment (UMHAT) Sveti Georgi, EAD - Clinic of Cardiology, Plovdiv
  - MHAT Dr. Bratan Shukjerov, Smolyan
  - Multiprofile Hospital For Active Treatment - Dr. Bratan Shukerov AD, Smolyan
  - Fifth Multiprofile Hospital for Active Treatment - Sofia EAD - Department of Cardiology, Sofia
  - Fifth Multiprofile Hospital for Active Treatment - Sofia EAD - Department of Endocrinology and Meteorism Diseases, Sofia
  - Medical Center Orfey OOD, Stara Zagora
- Czechia (8):
  - Lipidova poradna, Bílina
  - Medicus Services SRO, Brandýs nad Labem
  - Fakultni nemocnice Hradec Kralove, Klinika gerontologicka a metabolicka, Hradec Králové
  - Ordinace pro choroby srdce a cev, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
  - Oblastni nemocnice Trutnov, Oddeleni klinicke biochemie, Trutnov
  - MUDr. Nina Zemkova s.r.o. Interni Ambulance, Uherské Hradište
- Georgia (8):
  - Unimed Ajara LLC, Batumi
  - Clinic LJ Ltd, Kutaisi
  - Aleksandre Aladashvili Clinic - LLC, Tbilisi
  - Archangel St Michael Multiprofile Clinical Hospital Ltd, Tbilisi
  - Emergency Cardiology Center by Academician G. Chapidze Ltd, Tbilisi
  - Institute of Clinical Cardiology Ltd, Tbilisi
  - Unimed Kakheti - Caraps Medline LLC, Tbilisi
  - Unimed Kakheti - Telavi Referral Hospital LLC, Telavi
- Hungary (9):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - DRC Balatongyorok, Balatongyörök
  - Dr Lakatos Ferenc Belgyogyaszati-Kardiologiai Maganrendelo, Békéscsaba
  - Magyar Honvedseg Allami Egeszsegugyi Kozpont, II. sz Belgyogyaszat Osztaly, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - BKS Research Kft., Hatvan
  - Pecsi Tudomanyegyetem Klinikai Kozpont I.sz. Belgyogyaszati Klinika, Pécs
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Poland (12):
  - Indywidualna Specjalistyczna Praktyka Lekarska w Dziedzinie Kardiologii, lek. med. Krzysztof Cymerman, Gdynia
  - SALVIA Lekston i Madej s.j., Katowice
  - Malopolskie Centrum Alergii i Immunoterapii Allmedis SP Z O O, Krakow
  - AppleTreeClinics Sp. z o.o., Lodz
  - Nzoz Salusmed, Lodz
  - NZOZ All - Med Centrum Medyczne Specjalistyczne Gabinety Lekarskie Marcin Ogorek, Lodz
  - MEDICOME Sp. z o.o., Oświęcim
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Medyczne OMEGA SP Z O O, Płock
  - Clinmedica Research Omc Sp z o.o. Sp, Skierniewice
  - Centrum Kardiologiczne Pro Corde Sp. z o. o., Wroclaw
- Russia (41):
  - Northern Medical Clinical Center named after N.A. Semashko of the Federal Medical and Biological Agency, Arkhangelsk
  - First City Clinical Hospital n.a. E.E.Volosevich, Arkhangelsk
  - Altay Regional Cardiology Dispensary, Cardiology Department for Patients with Acute Myocardial Infarction, Barnaul
  - Chita State Medical Academy, Chita
  - Interregional Clinical Diagnostic Center, Kazan'
  - Kazan State Medical University based at City Clinical Hospital #7, Kazan'
  - Federal State Budget Institution "Scientific-Research Institute of Complex Problems of Cardiovascular Diseases, Kemerovo
  - Medical Center Alliance, Kirovsk
  - Krasnoyarsk State Medical University n.a. prof. V.F. Voino-Yasenetsky, Krasnoyarsk
  - National Medical Research Center of Preventive Medicine, Moscow
  - City Clinical Hospital #15 n.a. O.M. Filatov, Moscow
  - Central Clinical Hospital of Russian Academy of Sciences, Moscow
  - City Clinical Hospital n.a. M.E. Zhadkevich of Moscow Healthcare Department, Moscow
  - National Medical Research Center of Cardiology - Department of Atherosclerosis, Moscow
  - National Medical Research Center of Cardiology, Moscow
  - City Clinical Hospital n.a. M.P. Konchalovskiy, Moscow
  - Non-governmental Private Healthcare Institution "Scientific Clinical Centre of Open Joint-Stock Company Russian Railways" (JSC "RZD"), Moscow
  - Federal State Budget Institution "Outpatient Clinic #3" of Russian Federation President's Management Department, Moscow
  - City Clinical Hospital No.2, Novosibirsk
  - RC Medical LLC, Novosibirsk
  - Research Institute of Physiology and Fundamental Medicine, Novosibirsk
  - Orenburg State Medical University based at City Clinical Hospital #1, Orenburg
  - Clinical-diagnostic center Zdorovye, Rostov-on-Don
  - Rostov-on-Don City Hospital of Emergency Care, Rostov-on-Don
  - Clinic Complex JSC, Saint Petersburg
  - North-Western State Medical University named after I.I. Mechnikov, Saint Petersburg
  - Medical Technologies LLC, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Clinical Hospital #122 n. a. L.G. Sokolov of the Federal Medical Biological Agency, Saint Petersburg
  - Limited Liability Company MedPomosch, Saint Petersburg
  - City hospital #38 n.a. N.A. Semashko, Saint Petersburg
  - BioTechService LLC, Saint Petersburg
  - Consultative Diagnostic Center with Out-patient Clinic, Saint Petersburg
  - Almazov National Medical Research Centre, Scientific Laboratory of Electrocardiology, Saint Petersburg
  - Saint-Petersburg State Budget Healthcare Institution "City Pokrovskaya Hospital", Department of Cardiology N.3, Saint Petersburg
  - Regional Clinical Cardiology Dispensary, Saratov
  - Saratov State Medical University n. a. V.I. Razumovsky, Saratov
  - Tomsk National Research Medical Center of Russian Academy of Sciences, Tomsk
  - Autonomous Institution of healthcare of the Voronezh region "Voronezh regional clinical consultative and diagnostic centre, Voronezh
  - Yaroslavl Regional Clinical Hospital for War Veterans - International Center on the Problems of the Elderly "Zdorovoe Dolgoletie", Yaroslavl
  - Ural State Medical University based at Central City Clinical Hospital No.1 of Oktyabrskiy District, Yekaterinburg
- Ukraine (14):
  - Ivano-Frankivsk Regional Clinical Cardiological Dispensary, Chronic Ischaemic Heart Disease Department, Ivano-Frankivsk
  - Municipal Healthcare Institution Kharkiv City Clinical Hospital #27, Intensive Therapy Department, Kharkiv
  - Kharkiv Medical Academy of Postgraduate Education, Kharkiv
  - Kharkiv Railway Clinic. Hosp.#1, Branch Office of "Healthcare Center" of PJSC "Ukr. Railways", Cardiology Depart #2, Kharkiv
  - Kharkiv Railway Clinic. Hosp.#1, Branch Office of Healthcare Center of PJSC Ukr. Railways, Cardiology Depart #1, Kharkiv
  - Municipal Non-Commercial Enterprise "City Clinical Emergency Hospital n.a. prof. O.I. Meshchaninov of Kharkiv City Council, Kharkiv
  - Municipal Healthcare Institution Kharkiv City Outpatient Clinic #9, General Practice and Family Medicine Department #1, Kharkiv
  - Limited Liability Company Treatment and Diagnostic Center Adonis Plus, Outpatient Department, Kyiv
  - Kyiv City Clinical Hospital #1, Urgent Cardiology Department, Kyiv
  - SI Institute of Gerontology n.a. D.F.Chebotarev NAMS of Ukraine, Cardiol. Un. of Clin. Physiology and Int. Organs Path. Dep-t., Gen. Ther.Unit, Kyiv
  - SI Institute of Gerontology n.a. D.F.Chebotarev NAMS of Ukraine, Cardiol. Un. of Clin. Physiology and Int. Organs Path. Dep-t, Kyiv
  - Municipal Institution City Clinical Hospital #3 n.a. prof. L.J. Aleinikova, Cardiology Intensive Therapy Department, Odesa
  - Small Private Enterprise, Medical Centre Puls, Vinnytsia
  - Municipal Institution City Clinical Hospital #6, Therapeutic Department, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible patients entered a 4- to 6-week lifestyle stabilization period. The stabilization period was followed by a 2-week TG qualifying period, and patient eligibility was assessed based on the mean TG value from these 2 visits. If the patient's mean TG level during the TG qualifying period was ≥450 mg/dL (5.09 mmol/L) and <500 mg/dL (5.65 mmol/L), an additional TG measurement was taken 1 week later at Visit 3.1. The mean of all 3 TG measurements was used to determine eligibility for the study.
Groups:
- K-877: Participants randomized to receive K-877 0.2 mg tablets twice daily in the 12-week Efficacy Period continued to receive K-877 0.2 mg tablets BID in the 40-week Extension Period
- Placebo/Fenofibrate: Patients randomized to receive placebo matching K-877 0.2 mg BID in the 12-week Efficacy Period initiated fenofibrate dosing at 48 mg once daily at Visit 7 (Week 12). Starting from Visit 8 (Week 16), Investigators were allowed to adjust fenofibrate dosing (to 145 mg once daily) at their discretion according to the local standard of care.
Period: 12-week Efficacy
Arm/Group | K-877 | Placebo/Fenofibrate
Started (One participant was randomized but not assigned to a treatment group per physician decision.) | 311 | 159
Completed | 299 | 159
Not Completed | 12 | 0
Period: 40-week Extension
Arm/Group | K-877 | Placebo/Fenofibrate
Started (Note that 12 participants (7 participants in the K-877 group and 5 participants in the placebo/fenofibrate group) withdrew after completing the 12-week Efficacy Period and did not start the 40-week Extension Period.) | 292 | 154
Completed | 275 | 146
Not Completed | 17 | 8

BASELINE CHARACTERISTICS:
Population: One participant was randomized but not assigned to a treatment group per physician decision
Groups:
- K-877: K-877 0.2 mg Tablets
- Total: Total of all reporting groups
Arm/Group | K-877 | Placebo/Fenofibrate | Total
Number analyzed (Participants) | 311 | 159 | 470
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 220 | 119 | 339
  ≥65 years | 91 | 40 | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 40 | 134
  Male | 217 | 119 | 336
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 0 | 3
  Black or African American | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White | 302 | 157 | 459
  Other | 1 | 1 | 2
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 299 | 151 | 450
  Not reported/unknown | 0 | 1 | 1
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 793.44 (390.102) | 759.36 (395.359) | 781.45 (391.511)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Fasting TG From Baseline to Week 12
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Groups:
- Placebo: Placebo matching K-877 0.2 mg tablet BID
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -58.89 [-71.69 to -38.42] | -22.94 [-43.98 to 9.67]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

2. Secondary Outcome: Percent Change From Baseline to Week 12 in Remnant Cholesterol
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -55.51 [-71.29 to -33.64] | -13.29 [-43.30 to 9.76]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

3. Secondary Outcome: Percent Change From Baseline to Week 12 in HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 23.50 [5.24 to 45.13] | 7.33 [-4.00 to 18.79]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

4. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo A1
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 4.05 [-5.57 to 14.62] | 0.00 [-7.80 to 10.01]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0156, Hodges-Lehmann method

5. Secondary Outcome: Percent Change From Baseline to Week 12 in Non-HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -20.98 [-34.70 to -4.06] | -3.43 [-23.66 to 6.75]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

6. Secondary Outcome: Percent Change From Baseline to Week 12 in Total Cholesterol
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -14.55 [-25.74 to -1.19] | -2.05 [-17.59 to 7.37]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

7. Secondary Outcome: Percent Change From Baseline to Week 12 in LDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 31.49 [0.65 to 72.06] | 2.30 [-14.50 to 23.09]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

8. Secondary Outcome: Percent Change From Baseline to Week 12 in FFAs
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 303 | 154
Percent change | -25.25 [-48.37 to 3.74] | -5.51 [-32.64 to 28.65]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0001, Hodges-Lehmann method

9. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo A2
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 19.34 [7.27 to 35.41] | 0.00 [-8.09 to 6.38]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

10. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo B
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 0.57 [-14.90 to 16.66] | -1.67 [-11.71 to 12.54]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.5380, Hodges-Lehmann method

11. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo B48
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -36.64 [-71.42 to 17.61] | 19.91 [-18.96 to 101.41]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

12. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo B100
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 2.05 [-13.31 to 18.13] | -2.33 [-14.42 to 12.14]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.1165, Hodges-Lehmann method

13. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo C2
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -4.70 [-27.33 to 0.00] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0142, Hodges-Lehmann method

14. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo C3
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -41.97 [-54.44 to -21.64] | -3.10 [-25.16 to 18.08]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

15. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo E
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -29.09 [-44.73 to -6.92] | -5.98 [-28.29 to 12.15]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

16. Secondary Outcome: Change From Baseline to Week 12 in FGF21
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
pg/mL | 277.97 [37.31 to 650.73] | 12.15 [-162.80 to 112.46]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

17. Secondary Outcome: Change From Baseline to Week 12 in hsCRP
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
mg/L | -0.201 [-1.355 to 0.685] | -0.100 [-1.235 to 0.821]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.4589, Hodges-Lehmann method

18. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (VLDL Cholesterol-Large)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -36.45 [-55.39 to -5.31] | -5.95 [-27.52 to 30.89]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

19. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (VLDL Cholesterol-Intermediate)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -23.23 [-42.10 to 1.79] | 0.07 [-18.32 to 25.73]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

20. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (VLDL Cholesterol-Small)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -6.07 [-24.09 to 9.75] | 4.16 [-12.56 to 21.97]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Other; p < .0001, Hodges-Lehmann method

21. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Intermediate Density Lipoproteins 1)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -0.22 [-17.02 to 22.34] | 2.42 [-9.70 to 17.69]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.2486, Hodges-Lehmann method

22. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Intermediate Density Lipoproteins 2)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 17.52 [-2.00 to 39.87] | 3.21 [-9.58 to 17.69]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

23. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Low Density Lipoproteins I)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 44.20 [10.67 to 89.89] | 4.81 [-11.65 to 25.30]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

24. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Low Density Lipoproteins IIa)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 53.94 [14.68 to 112.53] | 4.24 [-16.31 to 23.16]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

25. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Low Density Lipoproteins IIb)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 48.44 [8.96 to 110.09] | 1.89 [-14.54 to 23.96]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

26. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Low Density Lipoproteins IIIa)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 23.79 [-19.17 to 76.61] | -0.80 [-13.28 to 17.39]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0001, Hodges-Lehmann method

27. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Low Density Lipoproteins IIIb)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -5.73 [-48.62 to 47.19] | 0.71 [-21.79 to 16.61]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.2763, Hodges-Lehmann method

28. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Low Density Lipoproteins IVa)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -30.48 [-59.53 to 7.01] | -2.89 [-20.28 to 16.04]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

29. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Low Density Lipoproteins IVb)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -35.08 [-54.14 to -15.21] | -0.74 [-21.22 to 19.16]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

30. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Low Density Lipoproteins IVc)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -23.39 [-38.34 to -11.75] | 0.89 [-15.75 to 15.88]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

31. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (High Density Lipoproteins 2b)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -10.65 [-19.15 to -0.88] | 0.91 [-9.59 to 11.60]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

32. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (High Density Lipoproteins 3 and 2a)
Description: Two lipoprotein subclasses, HDL3 and HDL2a, were analyzed together as one measurement without distinction.
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -2.13 [-10.90 to 7.50] | -0.53 [-8.50 to 9.19]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.1651, Hodges-Lehmann method

33. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility (Diameter of the Major LDL Particle (Å))
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | 2.67 [0.90 to 4.73] | 0.14 [-0.60 to 0.89]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

34. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction (VLDL & Chylomicron Particles)
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
Percent change | -42.76 [-61.49 to -15.41] | -5.59 [-29.00 to 24.71]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

35. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction (VLDL & Chylomicron Particles-Large)
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 12 Weeks
Population: Since there were one or multiple records with a baseline value of 0, the percent change cannot be determined for such records. In such cases, the secondary endpoints were evaluated for change from baseline to week 12.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
nmol/L | -12.62 [-31.63 to -3.27] | -3.75 [-18.37 to 8.30]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

36. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction (VLDL Particles-Medium)
Time Frame: 12 Weeks
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
nmol/L | -41.27 [-79.42 to -9.78] | -9.13 [-36.78 to 26.18]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

37. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction (VLDL Particles-Small)
Time Frame: 12 Weeks
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
nmol/L | 0.46 [-25.09 to 20.86] | 0.07 [-16.80 to 20.72]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.5107, Hodges-Lehmann method

38. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction (LDL Particles)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 309 | 159
Percent change | 17.58 [-13.32 to 60.38] | 4.97 [-15.42 to 25.30]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0018, Hodges-Lehmann method; Hodges-Lehmann method

39. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction (IDL Particles)
Time Frame: 12 Weeks
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
nmol/L | -17.06 [-123.66 to 39.24] | -2.74 [-87.30 to 76.76]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0742, Hodges-Lehmann method

40. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction (LDL Particles-Large)
Time Frame: 12 Weeks
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
nmol/L | 54.52 [0.00 to 306.49] | 0.00 [-13.04 to 43.85]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

41. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction (LDL Particles-Small)
Time Frame: 12 Weeks
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
nmol/L | 83.88 [-254.52 to 394.98] | 12.43 [-135.98 to 230.34]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.2707, Hodges-Lehmann method

42. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction (HDL Particles)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
Percent change | 5.96 [-8.43 to 23.02] | -1.60 [-13.63 to 11.21]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0009, Hodges-Lehmann method

43. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction (HDL Particles-Large)
Time Frame: 12 Weeks
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: µmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
µmol/L | 0.22 [-0.94 to 1.56] | 0.00 [-1.02 to 1.10]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.2879, Hodges-Lehmann method

44. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction (HDL Particles-Medium)
Time Frame: 12 Weeks
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: µmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
µmol/L | -0.21 [-3.98 to 2.90] | -0.23 [-2.96 to 1.66]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.9786, Hodges-Lehmann method

45. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction (HDL Particles-Small)
Time Frame: 12 Weeks
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: µmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
µmol/L | 1.54 [-2.95 to 7.78] | 0.16 [-4.19 to 4.35]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0075, Hodges-Lehmann method

46. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction (VLDL Particle Size)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
Percent change | -5.02 [-16.79 to 5.79] | -2.26 [-11.03 to 7.60]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0241, Hodges-Lehmann method

47. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction (LDL Particle Size)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 305 | 157
Percent change | 1.02 [0.00 to 3.54] | 0.00 [-0.53 to 0.54]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

48. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction (HDL Particle Size)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
Percent Change | -1.19 [-4.48 to 2.36] | -0.14 [-3.22 to 2.36]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0502, Hodges-Lehmann method

49. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction (Triglyceride)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
Percent change | -54.86 [-70.90 to -31.38] | -15.24 [-37.36 to 18.69]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

50. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction (VLDL & Chylomicron Triglyceride)
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 310 | 159
Percent change | -55.19 [-70.80 to -32.36] | -16.20 [-37.74 to 21.70]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

51. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction HDL Cholesterol (Total)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 305 | 154
Percent Change | 5.51 [-12.73 to 29.84] | -2.20 [-17.16 to 16.56]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0209, Hodges-Lehmann method

52. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of TG:HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -66.21 [-79.82 to -42.95] | -26.81 [-51.86 to 13.12]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

53. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of TC:HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -32.36 [-47.83 to -10.34] | -9.02 [-29.95 to 6.61]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

54. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of Non-HDL-C:HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -32.36 [-47.83 to -10.34] | -9.02 [-29.95 to 6.61]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

55. Secondary Outcome: Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of LDL-C:Apo B
Time Frame: 12 Weeks
Population: as for outcome 35
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Ratio | 0.219 [0.050 to 0.359] | 0.026 [-0.096 to 0.138]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, non-parametric Hodges-Lehmann method

56. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of Apo B:Apo A1
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -1.68 [-19.68 to 17.39] | -1.25 [-13.68 to 9.26]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0001, Hodges-Lehmann method

57. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of Apo C3:Apo C2
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 311 | 159
Percent change | -27.76 [-45.35 to -7.99] | -0.47 [-23.52 to 17.90]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

58. Secondary Outcome: Percent Change From Baseline to Week 52 in Fasting TG
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 146
Percent change | -59.96 [-74.38 to -41.52] | -49.55 [-64.80 to -26.83]

59. Secondary Outcome: Percent Change From Baseline to Week 52 in Remnant Cholesterol
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 269 | 145
Percent change | -58.39 [-72.45 to -39.62] | -43.31 [-60.66 to -24.59]

60. Secondary Outcome: Percent Change From Baseline to Week 52 in HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 146
Percent change | 18.78 [3.03 to 38.46] | 15.59 [5.26 to 32.35]

61. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo A1
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 143
Percent change | 3.29 [-6.51 to 12.10] | 2.56 [-6.62 to 12.31]

62. Secondary Outcome: Percent Change From Baseline to Week 52 in Non-HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 146
Percent change | -21.80 [-37.89 to -6.95] | -14.22 [-31.57 to 3.72]

63. Secondary Outcome: Percent Change From Baseline to Week 52 in TC
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 146
Percent change | -15.28 [-29.10 to -4.01] | -8.64 [-23.55 to 5.08]

64. Secondary Outcome: Percent Change From Baseline to Week 52 in LDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 269 | 145
Percent change | 31.90 [0.00 to 76.62] | 22.96 [1.41 to 51.68]

65. Secondary Outcome: Percent Change From Baseline to Week 52 in FFAs
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 219 | 127
Percent change | -21.61 [-46.76 to 8.15] | -21.41 [-45.70 to -1.02]

66. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo A2
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 143
Percent change | 15.92 [3.23 to 31.25] | 8.33 [0.00 to 20.69]

67. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo B
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 143
Percent change | -1.73 [-14.74 to 15.84] | 0.00 [-14.13 to 12.16]

68. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo B48
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 273 | 144
Percent change | -19.43 [-58.77 to 60.61] | -15.19 [-51.08 to 112.60]

69. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo B100
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 273 | 143
Percent change | -1.32 [-15.58 to 17.35] | -0.87 [-13.44 to 12.30]

70. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo C2
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 270 | 144
Percent change | -9.56 [-34.50 to 0.00] | 0.00 [-19.81 to 0.00]

71. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo C3
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 273 | 144
Percent change | -42.80 [-57.88 to -22.27] | -26.25 [-44.64 to -2.73]

72. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo E
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 143
Percent change | -30.82 [-49.25 to -13.04] | -30.00 [-42.59 to -9.76]

73. Secondary Outcome: Change From Baseline to Week 52 in FGF21
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 145
pg/mL | 371.80 [97.30 to 795.00] | 194.40 [57.00 to 524.10]

74. Secondary Outcome: Change From Baseline to Week 52 in hsCRP
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
mg/L | -0.100 [-1.400 to 0.900] | -0.225 [-1.700 to 0.750]

75. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (VLDL Cholesterol-Large)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | -36.60 [-57.18 to -9.94] | -22.03 [-46.31 to 3.89]

76. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (VLDL Cholesterol-Intermediate)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | -25.03 [-45.41 to -2.97] | -13.31 [-32.85 to 10.20]

77. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (VLDL Cholesterol-Small)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | -12.96 [-28.26 to 8.80] | -2.31 [-21.61 to 17.28]

78. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Intermediate Density Lipoproteins 1)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | 0.69 [-22.32 to 20.37] | 3.54 [-14.98 to 19.42]

79. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Intermediate Density Lipoproteins 2)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | 17.33 [-4.92 to 45.07] | 15.87 [-3.79 to 33.13]

80. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Low Density Lipoproteins I)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | 46.51 [11.45 to 96.51] | 25.53 [7.94 to 57.81]

81. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Low Density Lipoproteins IIa)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | 61.36 [18.02 to 121.43] | 33.66 [8.36 to 69.06]

82. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Low Density Lipoproteins IIb)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | 45.61 [10.19 to 110.03] | 27.29 [3.08 to 75.15]

83. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Low Density Lipoproteins IIIa)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | 18.50 [-17.32 to 76.72] | 19.64 [-9.16 to 55.84]

84. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Low Density Lipoproteins IIIb)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | -6.92 [-46.06 to 44.10] | 1.17 [-33.87 to 37.07]

85. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Low Density Lipoproteins IVa)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | -25.63 [-59.65 to 4.76] | -24.80 [-48.67 to 7.25]

86. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Low Density Lipoproteins IVb)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | -37.26 [-54.63 to -13.67] | -24.22 [-46.23 to -7.72]

87. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Low Density Lipoproteins IVc)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | -26.81 [-39.69 to -12.43] | -17.41 [-34.43 to -3.23]

88. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (High Density Lipoproteins 2b)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | -11.67 [-21.85 to -0.44] | -5.62 [-18.23 to 5.91]

89. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (High Density Lipoproteins 3 and 2a)
Description: Two lipoprotein subclasses, HDL3 and HDL2a, were analyzed together as one measurement without distinction.
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | -4.62 [-13.84 to 5.23] | -3.71 [-13.22 to 5.49]

90. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility (Diameter of the Major LDL Particle (Å))
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 144
Percent change | 2.69 [1.10 to 4.84] | 1.54 [0.71 to 3.24]

91. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction (VLDL & Chylomicron Particles)
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
Percent change | -40.10 [-63.62 to -14.91] | -28.98 [-48.61 to -2.98]

92. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction (VLDL & Chylomicron Particles-Large)
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 52 Weeks
Population: Since there were one or multiple records with a baseline value of 0, the percent change cannot be determined for such records. In such cases, the secondary endpoints were evaluated for change from baseline to week 52.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
nmol/L | -13.00 [-32.70 to -2.40] | -8.60 [-28.80 to -1.40]

93. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction (VLDL Particles-Medium)
Time Frame: 52 Weeks
Population: as for outcome 92
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
nmol/L | -41.95 [-77.20 to -5.10] | -26.90 [-64.80 to 4.80]

94. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction (VLDL Particles-Small)
Time Frame: 52 Weeks
Population: as for outcome 92
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
nmol/L | -0.15 [-18.10 to 19.60] | 0.00 [-16.60 to 24.70]

95. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction (LDL Particles)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
Percent change | 14.43 [-10.07 to 62.78] | 12.79 [-11.69 to 43.15]

96. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction (IDL Particles)
Time Frame: 52 Weeks
Population: as for outcome 92
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
nmol/L | -12.00 [-151.00 to 53.00] | -6.00 [-127.00 to 57.00]

97. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction (LDL Particles-Large)
Time Frame: 52 Weeks
Population: as for outcome 92
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
nmol/L | 53.00 [0.00 to 273.00] | 8.00 [0.00 to 199.00]

98. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction (LDL Particles-Small)
Time Frame: 52 Weeks
Population: as for outcome 92
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
nmol/L | 59.00 [-198.00 to 425.00] | 97.00 [-209.00 to 420.00]

99. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction (HDL Particles)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
Percent change | 4.96 [-9.59 to 20.58] | 0.00 [-9.74 to 13.49]

100. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction (HDL Particles-Large)
Time Frame: 52 Weeks
Population: as for outcome 92
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
umol/L | 0.20 [-0.90 to 1.50] | 0.30 [-1.10 to 1.70]

101. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction (HDL Particles-Medium)
Time Frame: 52 Weeks
Population: as for outcome 92
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
umol/L | -0.20 [-3.70 to 2.80] | -0.40 [-4.20 to 2.20]

102. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction (HDL Particles-Small)
Time Frame: 52 Weeks
Population: as for outcome 92
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
umol/L | 1.80 [-2.90 to 7.30] | 1.40 [-2.70 to 5.10]

103. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction (VLDL Particle Size)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
Percent change | -7.15 [-17.67 to 3.71] | -5.46 [-15.32 to 3.65]

104. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction (LDL Particle Size)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 237 | 131
Percent change | 1.03 [0.00 to 3.57] | 0.51 [-0.51 to 2.03]

105. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction (HDL Particle Size)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
Percent change | -1.14 [-4.35 to 2.27] | -1.15 [-4.35 to 1.15]

106. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction (Triglyceride)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
Percent change | -55.03 [-73.79 to -31.24] | -42.76 [-58.82 to -13.70]

107. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction (VLDL & Chylomicron Triglyceride)
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 258 | 137
Percent change | -54.30 [-73.74 to -30.73] | -41.55 [-58.97 to -17.39]

108. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction (HDL Cholesterol)
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 212 | 120
Percent change | 2.90 [-15.75 to 24.94] | -1.19 [-15.14 to 25.57]

109. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of TG:HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 146
Percent change | -66.38 [-81.70 to -45.55] | -56.61 [-71.34 to -32.09]

110. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of TC:HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 146
Percent change | -31.53 [-47.32 to -13.74] | -23.70 [-41.03 to -5.83]

111. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of Non-HDL-C:HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 146
Percent change | -36.49 [-53.81 to -16.78] | -27.67 [-47.17 to -7.02]

112. Secondary Outcome: Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of LDL-C:Apo B
Time Frame: 52 Weeks
Population: as for outcome 92
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 267 | 142
Ratio | 0.210 [0.050 to 0.420] | 0.150 [0.030 to 0.310]

113. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of Apo B:Apo A1
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 274 | 143
Percent change | -3.56 [-20.00 to 14.91] | -2.94 [-19.27 to 10.64]

114. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of Apo C3:Apo C2
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 270 | 144
Percent change | -27.81 [-43.96 to -4.95] | -13.17 [-32.52 to 4.21]

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Treatment-emergent adverse event (TEAE) was defined as any adverse event that occurred for the first time after the first dose of double-blind study drug or existed prior to the first dose and worsened during the post-dosing period.
Groups:
- K-877: 12-Week Efficacy: * K-877 0.2 mg Tablets BID
  * Only AEs with onset in the 12-week efficacy period are included.
- Placebo:12-Week Efficacy: * Placebo matching K-877 0.2 mg BID
  * Only AEs with onset in the 12-week efficacy period are included.
- K-877: 40-Week Extension: * Participants randomized to receive K-877 0.2 mg tablets twice daily in the 12-week Efficacy Period continued to receive K-877 0.2 mg tablets BID in the 40-week Extension Period
  * Only AEs with onset in the 40-week extension period are included.
- Fenofibrate 40-Week Extension: * Patients randomized to receive placebo matching K-877 0.2 mg BID in the 12-week Efficacy Period initiated fenofibrate dosing at 48 mg once daily at Visit 7 (Week 12). Starting from Visit 8 (Week 16), Investigators were allowed to adjust fenofibrate dosing (to 145 mg once daily) at their discretion according to the local standard of care.
  * Only AEs with onset in the 40-week extension period are included.
Arm/Group | K-877: 12-Week Efficacy | Placebo:12-Week Efficacy | K-877: 40-Week Extension | Fenofibrate 40-Week Extension
All-Cause Mortality (participants affected / at risk) | 3/311 | 0/159 | 3/292 | 1/154
Serious Adverse Events (participants affected / at risk) | 11/311 | 3/159 | 25/292 | 5/154
Other Adverse Events (participants affected / at risk) | 0/311 | 0/159 | 2/292 | 8/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | K-877: 12-Week Efficacy (N=311) | Placebo:12-Week Efficacy (N=159) | K-877: 40-Week Extension (N=292) | Fenofibrate 40-Week Extension (N=154)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Endometritis (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 3 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | K-877: 12-Week Efficacy (N=311) | Placebo:12-Week Efficacy (N=159) | K-877: 40-Week Extension (N=292) | Fenofibrate 40-Week Extension (N=154)
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (5):
  • Study Protocol: Ver.1.0 (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT03011450/Prot_000.pdf
  • Study Protocol: Ver.2.0 (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT03011450/Prot_001.pdf
  • Statistical Analysis Plan: V1.0 (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03011450/SAP_002.pdf
  • Statistical Analysis Plan: V2.0 (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03011450/SAP_003.pdf
  • Statistical Analysis Plan: Addendum (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03011450/SAP_004.pdf